CLINICAL TRIAL: NCT02097017
Title: Prophylactic Lidocaine Spray for Pain Alleviation in Women Undergoing Osmotic Dilator Insertion for Second Trimester Dilatation and Evacuation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Dr. Avi Shina MD, Doctor, Sheba Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SHEBA-14-0801-AS-CTIL
Record Dates: First submitted 2014-03-23; First posted 2014-03-26 (Estimated); Last update posted 2020-05-27 (Actual); Status verified 2020-05

CONDITIONS: Pain Alleviation; Dilatation and Evacuation; Laminaria Placement
Keywords: lidocaine; laminaria; dilatation and evacuation; pain
MeSH Terms: conditions — Dilatation, Pathologic; Pain | interventions — Lidocaine

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- lidocaine spray group (Active Comparator)
  Interventions: Drug: Lidocaine
- placebo arm (Placebo Comparator)
  Interventions: Other: placebo comparator

INTERVENTIONS:
Drug: Lidocaine — will local application of lidocaine to the cervix alleviate pain of laminaria insertion
  Arms: lidocaine spray group
Other: placebo comparator
  Arms: placebo arm

SUMMARY:
To examine whether application of lidocaine spray in cervical preparation for second trimester dilatation and evacuation alleviates pain and is superior to current protocol of preparation without analgesia and superior to placebo.

a double- blind, randomized, placebo- controlled trial, performed at a single tertiary medical center. Eligible participants aged 18 and older and about to undergo dilation & evacuation of the uterus between 12 to 24 weeks of gestation. Participants will be randomized using computer generated allocation to receive 10% Xylocaine (lidocaine group) spray or normal saline 0.9% (placebo group), applied identically topically to the endocervix and ectocervix before laminaria insertion. The primary outcome will be the participant's reported pain score immediately after the first laminaria was inserted as measured on a 10 cm visual analog scale (VAS). Secondary outcomes wiil be reported pain scores at speculum removal, 15 minutes after speculum insertion and immediately before the D&E procedure.

ELIGIBILITY:
Inclusion Criteria:

* • Informed consent

  * Women with a gestational age of 12-24 weeks by last menstrual period.

Exclusion Criteria:

* • CRL assesed by ultrasound as <10 weeks

  * Clinical Uterine size >24 weeks
  * Fetus Bi Parietal Diameter > 50 mm
  * Known amide allergy

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 134 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2018-08-01 (Actual); Study Completion 2018-08-01 (Actual)

PRIMARY OUTCOMES:
Pain immediately after inserton of first laminaria | immediately after first laminaria insertion
  Women's reported VAS pain score immediately after the insertion of the first laminaria.

SECONDARY OUTCOMES:
Reported pain afer speculum removal, 15 minutes after speculum inserion and before D&E | After speculum removal, 15 minutes after speculum insertion and before D&E
  Reported VAS pain at speculum removal, 15 minutes after speculum insertion and before D&E

CONTACTS AND LOCATIONS:
Locations (1):
- Sheba Medical Center, Ramat Gan, Israel